CLINICAL TRIAL: NCT00823212
Title: PLATINUM: A Prospective, Randomized, Multicenter Trial to Assess an Everolimus-Eluting Coronary Stent System (PROMUS Element™) for the Treatment of up to Two De Novo Coronary Artery Lesions
Brief Title: The PLATINUM Clinical Trial to Assess the PROMUS Element Stent System for Treatment of De Novo Coronary Artery Lesions
Acronym: PLATINUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2046; ACTRN12608000582358
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stents; DES; atherosclerotic
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; thienopyridine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PROMUS (Active Comparator): Patients who received the PROMUS (XIENCE V) Everolimus-Eluting Coronary Stent
  Interventions: Device: PROMUS Coronary Stent System; Drug: Aspirin; Drug: Thienopyridine
- PROMUS Element (Experimental): Patients who received the PROMUS™ Element Everolimus-Eluting Coronary Stent
  Interventions: Device: PROMUS Element Coronary Stent System; Drug: Aspirin; Drug: Thienopyridine

INTERVENTIONS:
Device: PROMUS Coronary Stent System — PROMUS is a device/drug combination product composed of two components, a device (coronary stent system including a cobalt chromium stent platform) and a drug product (a formulation of everolimus contained in a polymer coating).
  Other Names: XIENCE V
  Arms: PROMUS
Device: PROMUS Element Coronary Stent System — PROMUS Element is a device/drug combination product composed of two components, a device (coronary stent system including a platinum chromium stent platform) and a drug product (a formulation of everolimus contained in a polymer coating that is the same as on the PROMUS [XIENCE V] stent).
  Arms: PROMUS Element
Drug: Aspirin — Patients are required to take aspirin indefinitely after stent implant. It is recommended that aspirin 162-325 mg daily be given for at least 6 months after stent placement and that aspirin 75-162 mg daily be given indefinitely thereafter.
Drug: Thienopyridine — Patients must be treated with one of the following thienopyridines for at least 6 months following the index procedure: clopidogrel 75 mg daily; or ticlopidine 250 mg twice daily; or prasugrel (outside the United States and if approved at the time of the procedure). If used, the prescribed dose should be in accordance with approved country-specific labeling. In patients not at high risk of bleeding, thienopyridine treatment should continue for at least 12 months after stent implant.
  Other Names: A brand name for clopidogrel is PLAVIX.; A brand name for ticlopidine is TICLID.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the PROMUS Element™ Everolimus-Eluting Coronary Stent System for the treatment of patients with up to 2 de novo atherosclerotic coronary artery lesions.

This clinical trial compares outcomes in patients treated with PROMUS Element to those in patients treated with a different everolimus-eluting coronary stent. The lesions are of average length in average-sized vessels ("workhorse"). A companion sub-trial evaluates outcomes in smaller vessels (SV) and another sub-trial evaluates outcomes in longer lesions (LL).

DETAILED DESCRIPTION:
The wide-spread use of DES has evolved as standard of care in de novo lesions. The proposed study will evaluate the safety and effectiveness of PROMUS Element for the treatment of de novo atherosclerotic lesions in native coronary arteries. The study design is consistent with the draft guidance for industry titled, "Coronary Drug-Eluting Stents - Nonclinical and Clinical Studies" (March 2008).

During the trial, thienopyridines must be administered according to the 2007 American College of Cardiology (ACC)/American Heart Association (AHA)/Society for Cardiovascular Angiography and Interventions (SCAI) guidelines, which recommended that clopidogrel (75 mg daily) or ticlopidine (250 mg twice daily) be prescribed after stent implantation for at least 6 months in all patients, and for at least 12 months in patients who are not at high risk of bleeding. For sites in the United States, the use of prasugrel is not allowed as part of the PLATINUM Clinical Trial. For sites in other countries, prasugrel may be prescribed according to its approved dosing in countries in which it is available. For patients taking aspirin daily a loading dose is recommended; for patients who have not been taking aspirin daily, aspirin must be administered as a loading dose. Patients continue to take aspirin indefinitely to reduce the risk of thrombosis.

The main study is the PLATINUM Workhorse Randomized Controlled Trial, which is registered under NCT00823212. The clinical protocol includes two companion sub-trials with smaller vessels (PLATINUM SV) and longer lesions (PLATINUM LL) plus a Pharmacokinetics sub-trial (PLATINUM PK). The three sub-trials are registered under separate NCT numbers.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient (or legal guardian) understands study requirements and treatment procedures and provides written informed consent before any study-specific tests or procedures are performed
* For patients less than 20 years of age enrolled at a Japanese site, patient and patient's legal representative must provide written informed consent before any study-specific tests or procedures are performed
* Patient is eligible for percutaneous coronary intervention (PCI)
* Patient has documented stable angina pectoris or documented silent ischemia; or unstable angina pectoris
* Patient is an acceptable candidate for coronary artery bypass grafting (CABG)
* Patient has a left ventricular ejection fraction (LVEF) >=30% as measured within 30 days prior to enrollment
* Patient is willing to comply with all protocol-required follow-up evaluations

Angiographic Inclusion Criteria (visual estimate):

- Target lesion must be a de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter (RVD) >=2.50 mm and <=4.25 mm. Target lesion length must measure (by visual estimate) <=24 mm. Target lesion must be in a major coronary artery or branch with visually estimated stenosis >=50% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow >1.

Exclusion Criteria:

* Patient has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute myocardial infarction (MI)
* Patient has had a known diagnosis of recent MI (ie, within 72 hours prior to index procedure) and has elevated enzymes at time of index procedure as follows.

  * Patients are excluded if any of the following criteria are met at time of the index procedure.

    * If creatine kinase-myoglobin band (CK-MB) >2× upper limit of normal (ULN), the patient is excluded regardless of CK Total.
    * If CK-MB is 1-2× ULN, the patient is excluded if the CK Total is >2× ULN.
  * If CK Total/CK MB are not used and Troponin is, patients are excluded if the following criterion is met at time of index procedure.

    * Troponin >1× ULN with at least one of the following.

      * Patient has ischemic symptoms and ECG changes indicative of ongoing ischemia (eg, >1 mm ST segment elevation or depression in consecutive leads or new left bundle branch block [LBBB]);
      * Development of pathological Q waves in the ECG; or
      * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

Note: For patients with unstable angina or patients who have had a recent MI, CK Total/CK MB (or Troponin if CK Total/CK MB are not used) must be documented prior to enrolling/randomizing the patient.

* Patient has received an organ transplant or is on a waiting list for an organ transplant
* Patient is receiving or scheduled to receive chemotherapy within 30 days before or after index procedure
* Patient is receiving oral or intravenous immunosuppressive therapy (ie, inhaled steroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (eg, human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
* Patient is receiving chronic (>=72 hours) anticoagulation therapy (eg, heparin, coumadin) for indications other than acute coronary syndrome
* Patient has platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Patient has white blood cell (WBC) count <3,000 cells/mm3
* Patient has documented or suspected liver disease, including laboratory evidence of hepatitis
* Patient is on dialysis or has known renal insufficiency (ie, estimated creatinine clearance <50 ml/min by the Cockcroft Gault formula, or [(140-age)*lean body weight (in kg)]/[plasma creatinine (mg/dl)*72])
* Patient has history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Target vessel(s) or side branch has been treated with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to index procedure
* Target vessel(s) has been treated within 10 mm proximal or distal to target lesion (by visual estimate) with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) at any time prior to index procedure
* Non-target vessel or side branch has been treated with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 24 hours prior to index procedure
* Planned or actual target vessel(s) treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter immediately prior to stent placement
* Planned PCI or CABG after index procedure
* Patient previously treated at any time with coronary intravascular brachytherapy
* Patient has a known allergy to the study stent system or protocol-required concomitant medications (eg, stainless steel, platinum, cobalt, chromium, nickel, tungsten, acrylic, fluoropolymers, everolimus, thienopyridines, aspirin, contrast) that cannot be adequately premedicated
* Patient has active peptic ulcer or active gastrointestinal (GI) bleeding
* Patient has one of the following.

  * Other serious medical illness (eg, cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
  * Current problems with substance abuse (eg, alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with protocol or confound data interpretation
* Patient is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Patient intends to participate in another investigational drug or device clinical trial within 12 months after index procedure
* Patient with known intention to procreate within 12 months after index procedure (Women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure.)
* Patient is a woman who is pregnant or nursing (A pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
* Patient has more than 2 target lesions, or more than 1 target lesion and 1 non-target lesion, which will be treated during the index procedure

Angiographic Exclusion Criteria (visual estimate):

* Target lesion meets any of the following criteria:

  * Aorto-ostial location (ie, lesion located within 5 mm of ostium by visual estimate)
  * Left main location
  * Located within 5 mm of origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery by visual estimate
  * Located within a saphenous vein graft or arterial graft
  * Will be accessed via a saphenous vein graft or arterial graft
  * Involves a side branch >=2.0 mm in diameter by visual estimate
  * Involves a clinically significant side branch <2.0 mm in diameter by visual estimate that has a clinically significant stenosis at the ostium
  * TIMI flow 0 (total occlusion) or TIMI flow 1 prior to wire crossing
  * Excessive tortuosity proximal to or within the lesion
  * Extreme angulation proximal to or within the lesion
  * Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified by visual estimate
  * Restenotic from previous intervention
  * Thrombus, or possible thrombus, present in target vessel
* Non-target lesion to be treated during the index procedure meets any of the following criteria:

  * Located within the target vessel
  * Located within a bypass graft (venous or arterial)
  * Left main location
  * Chronic total occlusion
  * Involves a complex bifurcation (eg, bifurcations requiring treatment with more than 1 stent)
  * Restenotic from previous intervention
* Patient has unprotected left main coronary artery disease (>50% diameter stenosis)
* Patient has protected left main coronary artery disease and a target lesion in the LAD or LCX
* Patient has an additional clinically significant lesion(s) in target vessel for which an intervention within 12 months after the index procedure is likely to be required
* Patient has 2 target lesions in the same vessel that are separated by less than 15 mm (by visual estimate) Note: Multiple focal stenoses will be considered as a single lesion if they can be completely covered with 1 stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1530 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (133):
- United States (75):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Banner Good Samaritan Regional Medical Center, Phoenix, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Scripps Clinic, La Jolla, California
  - Good Samaritan Hospital, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - University of California San Diego, San Diego, California
  - Alvarado Hospital, San Diego, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Medical Center of the Rockies (Loveland), Loveland, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - MediQuest Research Group Inc. at Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - Southern Illinois University Memorial Medical Center, Springfield, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - Jewish Hospital and St. Mary's Healthcare, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic Foundation, Rochester, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital / Mid America Heart Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Kaleida Health, Buffalo, New York
  - Mount Sinai School Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Moses H. Cone Memorial Hospital/LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Ohio Health Research and Innovation Institute, Columbus, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Trinity Mother Frances Health System, Tyler, Texas
  - Lynchburg General Hospital, Lynchburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Providence Health & Services - Washington, Spokane, Washington
  - Aspirus Heart and Vascular Institute - Research and Education, Wausau, Wisconsin
- Australia (4):
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Royal Perth Hospital, Perth
  - The Prince Charles Hospital, Queensland
- Allgemeines Krankenhauas AKH, Vienna, Austria
- Belgium (4):
  - Academisch Ziekenhuis Middelheim, Antwerp
  - Ziekenhuis Oost Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Gasthuisberg, Leuven
- Denmark (2):
  - Skejby Sygehus, Aarhus
  - Rigshospitalet Copenhagen, Copenhagen
- Finland (3):
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (6):
  - CHU de Besancon, Besançon
  - Clinique St. Augustin, Bordeaux
  - Institut Cardiovasculaire - Paris Sud / Institut Hospitalier Jacques Cartier, Massy
  - Clinique du Millenaire, Montpellier
  - Centre Hopital Universitaire Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (6):
  - Kerckhoff Klinik, Bad Nauheim
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH, Bad Segeberg
  - Universitatsklinik Charite Berlin, Berlin
  - Universitat Heidelberg, Heidelberg
  - Herzzentrum Universitat Leipzig, Leipzig
- Japan (10):
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Japan Community Health Care Organization Hokkaido Hospital, Sapporo, Hokkaido
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Saiseikai Yokohama-City Eastern Hospital, Yokohama, Kanagawa
  - Sakakibara Heart Institute, Japan Research Promotion Society for Cardiovascular Diseases, Fuchu-shi, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - The Cardiovascular Institute Hospital, Minato-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Sakurabashi Watanabe Hospital, Osaka
- P. Stradins University Hospital, Riga, Latvia
- Malaysia (2):
  - Sarawak General Hospital, Kota Samarahan, Sarawak
  - Institut Jantung Negara, Kuala Lumpur
- Netherlands (4):
  - Medisch Centrum Alkmaar, Alkmaar
  - Amphia Ziekenhuis, Breda
  - Catherina Ziekenhuis, Eindhoven
  - St Antonius Ziekenhuis, Nieuwegein
- New Zealand (3):
  - Middlemore Hospital, Otahuhu, Auckland
  - Ascot Angiography, Auckland
  - Wellington Hospital, Wellington
- Poland (4):
  - Szpital Uniwersytecki, Bydgoszcz
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - National Institute of Cardiology, Warsaw
  - Military Hospital, Wroclaw
- Hospital De Santa Cruz, Carnaxide, Portugal
- National Heart Centre Singapore, Singapore, Singapore
- United Kingdom (6):
  - Guys and St. Thomas NHS Foundation Trust St. Thomas Hospital, London, England
  - James Cook University Hospital, Middlesbrough, England
  - John Radcliffe Infirmary Oxford II, Oxford, England
  - Royal Victoria Hospital, Belfast, Ireland
  - Golden Jubilee National Hospital, Clydebank
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

REFERENCES:
- [Result] Stone GW, Teirstein PS, Meredith IT, Farah B, Dubois CL, Feldman RL, Dens J, Hagiwara N, Allocco DJ, Dawkins KD; PLATINUM Trial Investigators. A prospective, randomized evaluation of a novel everolimus-eluting coronary stent: the PLATINUM (a Prospective, Randomized, Multicenter Trial to Assess an Everolimus-Eluting Coronary Stent System [PROMUS Element] for the Treatment of Up to Two de Novo Coronary Artery Lesions) trial. J Am Coll Cardiol. 2011 Apr 19;57(16):1700-8. doi: 10.1016/j.jacc.2011.02.016. Epub 2011 Apr 4. PMID 21470815
- [Derived] Kelly CR, Teirstein PS, Meredith IT, Farah B, Dubois CL, Feldman RL, Dens J, Hagiwara N, Rabinowitz A, Carrie D, Pompili V, Bouchard A, Saito S, Allocco DJ, Dawkins KD, Stone GW. Long-Term Safety and Efficacy of Platinum Chromium Everolimus-Eluting Stents in Coronary Artery Disease: 5-Year Results From the PLATINUM Trial. JACC Cardiovasc Interv. 2017 Dec 11;10(23):2392-2400. doi: 10.1016/j.jcin.2017.06.070. PMID 29217001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of 1,532 patients was planned; 1,530 patients (762 PROMUS and 768 PROMUS Element) were enrolled and randomized at 132 clinical sites from January 27, 2009 to September 4, 2009. Of these, 788 patients were from the USA, 562 from Europe, 124 from Japan, and 56 from the Asia-Pacific region excluding Japan.
Groups:
- PROMUS: Participants randomized to treatment with PROMUS everolimus-eluting stent (control device)
- PROMUS Element: Participants randomized to treatment with PROMUS Element everolimus-eluting stent (investigational device)
Period: Overall Study
Arm/Group | PROMUS | PROMUS Element
Started | 762 | 768
Completed | 727 (12-month follow-up) | 735 (12-month follow-up)
Not Completed | 35 | 33
Not completed — Death | 8 | 10
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Incarcerated | 0 | 1
Not completed — Missed 12-month visit | 21 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROMUS | PROMUS Element | Total
Number analyzed (Participants) | 762 | 768 | 1530
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 413 | 377 | 790
  >=65 years | 349 | 391 | 740
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.11 (10.28) | 63.99 (10.27) | 63.55 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 218 | 438
  Male | 542 | 550 | 1092
Race/Ethnicity, Customized [Number; unit: participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participant
    Caucasian | 644 | 650 | 1294
    Hispanic or Latino | 15 | 13 | 28
    Asian | 68 | 75 | 143
    Black of African heritage | 21 | 18 | 39
    Native Hawaiian or other Pacific Islander | 4 | 3 | 7
    American Indian or Alaska Native | 4 | 3 | 7
    Other | 1 | 4 | 5
    Maori | 0 | 1 | 1
    Not Disclosed | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 396 | 392 | 788
  Japan | 61 | 63 | 124
  Europe | 276 | 286 | 562
  Pacifica | 29 | 27 | 56
Cardiac History [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    Previous Percutaneous Coronary Intervention (PCI) | 247 | 238 | 485
    Previous Coronary Artery Bypass Graft (CABG) | 40 | 45 | 85
    Previous Myocardial Infarction (MI) | 160 | 160 | 320
    Congestive Heart Failure | 50 | 57 | 107
    Stable Angina | 463 | 474 | 937
    Unstable Angina | 188 | 185 | 373
    Silent Ischemia | 143 | 128 | 271
Cardiac History-Ejection Fraction [Mean (Standard Deviation); unit: Percent Ejection Fraction] | 59.04 (9.54) | 59.53 (10.07) | 59.29 (9.81)
Cardiac Risk Factor [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    Smoking, Ever | 448 | 493 | 941
    Medically Treated Diabetes | 191 | 169 | 360
    Hyperlipidemia Requiring Medication | 579 | 598 | 1177
    Hypertension Requiring Medication | 558 | 544 | 1102
    Family History of Coronary Artery Disease | 401 | 392 | 793
Comorbidities [Number; unit: Participants] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participants
    History of Peripheral Vascular Disease | 66 | 70 | 136
    History of Transient Ischemic Attack | 13 | 31 | 44
    History of Cerebrovascular Accident | 23 | 27 | 50
    History of Renal Disease | 23 | 26 | 49
    History of Gastrointestinal Bleeding | 8 | 10 | 18
Lesion Characteristic: Target Lesion Vessel [Number; unit: Lesion] — Reported per lesion. The same participant may have been treated for >1 lesion and therefore may be included in more than one category. Thus, the total number of lesions for this baseline measure does not equal the total number of participants in the group.
  Lesion
    Left Anterior Descending Artery | 354 | 357 | 711
    Left Circumflex Artery | 219 | 222 | 441
    Right Coronary Artery | 268 | 273 | 541
Lesion Characteristic: Lesion Location [Number; unit: Lesions] — Reported per lesion. The same participant may have been treated for >1 lesion and therefore may be included in more than one category. Thus, the total number of lesions for this baseline measure does not equal the total number of participants in the group.
  Lesions
    Ostial | 30 | 33 | 63
    Proximal | 338 | 348 | 686
    Mid | 401 | 387 | 788
    Distal | 72 | 84 | 156
Lesion Characteristics [Mean (Standard Deviation); unit: Millimeters]
  Reference Vessel Diameter | 2.63 (0.49) | 2.67 (0.49) | 2.65 (0.49)
  Minimum Lumen Diameter | 0.74 (0.34) | 0.75 (0.35) | 0.75 (0.34)
  Lesion Length | 12.50 (5.51) | 12.95 (5.74) | 12.72 (5.63)
Lesion Characteristic-Percent Diameter Stenosis [Mean (Standard Deviation); unit: Percent Diameter Stenosis] | 71.90 (11.47) | 71.81 (11.46) | 71.86 (11.46)
Lesion Characteristics [Number; unit: Lesions] — Reported per lesion. The same participant may have been treated for >1 lesion and therefore may be included in more than one category. Thus, the total number of lesions for this baseline measure does not equal the total number of participants in the group.
  Lesions
    Eccentric Lesion | 454 | 477 | 931
    > 45 Degree Bend | 142 | 148 | 290
    > 90 Degree Bend | 18 | 13 | 31
    Tortuosity, any | 62 | 72 | 134
    Calcification, any | 236 | 238 | 474
    Total Occlusion | 6 | 5 | 11
    Bifurcation | 62 | 78 | 140
Lesion Characteristics: American College of Cardiology (ACC)/American Heart Association (AHA) Class [Number; unit: Lesions] — Type A: minimally complex, readily accessible, non-angulated, smooth contour, little to no calcification, less than totally occlusive, not ostial in location, no major side branch involvement, absence of thrombus.
  Type B: moderately complex, eccentric, moderate tortuosity and angulation, moderate or heavy calcification, total occlusion < 3 months old, ostial location with presence of thrombus.
  Type C: severely complex, diffuse, excessive tortuosity and angulation, total occlusions > 3 months old, degenerated vein grafts,friable lesions
  Lesions
    Type A | 82 | 72 | 154
    Type B1 | 225 | 223 | 448
    Type B2 | 361 | 378 | 739
    Type C | 173 | 179 | 352
Lesion Characteristic - Pre-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: Lesion] — TIMI 0 - No perfusion TIMI 1 - Penetration with minimal perfusion TIMI 2 - Partial perfusion TIMI 3 - Complete perfusion A participant may be treated for >1 lesion, therefore the number of lesions for this baseline measure does not equal the total number of participants in the group.
  Lesion
    TIMI 0 | 0 | 0 | 0
    TIMI 1 | 6 | 5 | 11
    TIMI 2 | 27 | 29 | 56
    TIMI 3 | 808 | 818 | 1626

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure (TLF)
Description: Defined as any ischemia-driven revascularization of the target lesion, myocardial infarction (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel.
Time Frame: 12-month post index procedure
Population: The primary analysis set for the non-inferiority testing of the primary endpoint, 12-month TLF, is the per-protocol analysis set. All randomized participants who received their assigned treatment are included in the per-protocol analysis set.
Measure: Number; unit: percentage of participants
Groups:
- PROMUS: PROMUS everolimus-eluting stent (EES) implanted using standard percutaneous coronary intervention (PCI) technique
- PROMUS Element: PROMUS Element everolimus-eluting stent (EES) implanted using standard percutaneous coronary intervention (PCI) technique
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 714 | 731
percentage of participants | 2.9 | 3.4
Statistical Analysis 1: Comparison: PROMUS vs PROMUS Element; Study had 89% statistical power to demonstrate non-inferiority for target lesion failure (TLF, accounting for an expected 1-year attrition rate of 5%), assuming a 1-year TLF rate of 5.5% for both stents; Test type: Non-Inferiority or Equivalence — A 2-group Farrington-Manning test was used to test the 1-sided hypothesis of non-inferiority in differences with a non-inferiority margin of 3.5%. A p value <0.05 would indicate non-inferiority and correspond to the upper limit of the 1-sided 95% confidence interval of the difference not exceeding 3.5%; p = 0.001, Farrington-Manning test; Difference in percent of participants = 0.5, 95% CI 1-sided [upper limit 2.13] — The standard error for the difference was estimated according to the Farrington-Manning test

2. Secondary Outcome: Target Lesion Failure (TLF)
Description: TLF is defined as any ischemia-driven revascularization of the target lesion, myocardial infarction (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel.
Time Frame: 30 days
Population: Analysis was intention to treat; all patients in the study underwent clinical follow up to provide the information needed for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
Percentage of participants | 1.4 | 0.9

3. Secondary Outcome: Target Lesion Failure (TLF)
Description: as for outcome 2
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 756 | 763
percentage of participants | 1.9 | 1.7

4. Secondary Outcome: Target Lesion Failure (TLF)
Description: as for outcome 2
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 727 | 742
percentage of participants | 3.2 | 3.5

5. Secondary Outcome: Target Vessel Failure (TVF)
Description: TVF is defined as any ischemia-driven revascularization of the target vessel, MI (Q-wave and non-Q-wave) related to the target vessel or death related to the target vessel. For the purposes of this protocol, if it cannot be determined with certainty whether the MI or death was related to the target vessel, it will be considered a TVF.
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 1.4 | 0.9

6. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 5
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 756 | 763
percentage of participants | 2.0 | 1.8

7. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 5
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 727 | 742
percentage of participants | 4.0 | 4.2

8. Secondary Outcome: Myocardial Infarction (MI) Related to the Target Vessel
Description: Development of new Q-waves in ≥2 leads lasting ≥0.04 seconds with CK-MB/troponin levels above normal; if no new Q-waves, total creatine kinase (CK) >3x normal (peri-percutaneous coronary intervention [PCI]) or >2x normal (spontaneous) with elevated CK-MB, or troponin >3x normal (peri-PCI) or >2x normal (spontaneous) plus one of the following: ECG changes indicating new ischemia (new ST-T changes/left bundle branch block), imaging evidence of new loss of viable myocardium, new regional wall motion abnormality. Similar criteria for MI post bypass graft surgery, with CK-MB or troponin >5x normal
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 1.3 | 0.7

9. Secondary Outcome: Myocardial Infarction (MI) Related to the Target Vessel
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 1.4 | 0.7

10. Secondary Outcome: Myocardial Infarction (MI) Related to the Target Vessel
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 1.4 | 0.7

11. Secondary Outcome: All Cause Mortality
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of patients | 0.1 | 0.1

12. Secondary Outcome: All Cause Mortality
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 0.5 | 0.8

13. Secondary Outcome: All Cause Mortality
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 1.2 | 1.3

14. Secondary Outcome: Cardiac Death Related to the Target Vessel
Description: Cardiac death is defined as Death due to any of the following: acute myocardial infarction (MI); cardiac perforation/pericardial tamponade; arrhythmia or conduction abnormality; cerebrovascular accident (CVA) through hospital discharge or CVA suspected of being related to the procedure; complication of the procedure including bleeding, vascular repair, transfusion reaction, or bypass surgery or any death in which a cardiac cause cannot be excluded
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 0.0 | 0.1

15. Secondary Outcome: Cardiac Death Related to the Target Vessel
Description: as for outcome 14
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 0.1 | 0.5

16. Secondary Outcome: Cardiac Death Related to the Target Vessel
Description: as for outcome 14
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 0.4 | 0.8

17. Secondary Outcome: Non-cardiac Death
Description: Defined as a death not due to cardiac causes (see definition of cardiac death above)
Time Frame: 30 Days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 0.0 | 0.0

18. Secondary Outcome: Non-cardiac Death
Description: Defined as a death not due to cardiac causes (see definition of cardiac death above)
Time Frame: 6 Months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 0.1 | 0.3

19. Secondary Outcome: Non-cardiac Death
Description: Defined as a death not due to cardiac causes (see definition of cardiac death above)
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 0.5 | 0.4

20. Secondary Outcome: Cardiac Death or Myocardial Infarction (MI)
Description: Cardiac death is defined as death due to any of the following: acute myocardial infarction (MI); cardiac perforation/pericardial tamponade; arrhythmia or conduction abnormality; cerebrovascular accident (CVA) through hospital discharge or CVA suspected of being related to the procedure; complication of the procedure including bleeding, vascular repair, transfusion reaction, or bypass surgery or any death in which a cardiac cause cannot be excluded; see definition of MI above
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 1.4 | 0.8

21. Secondary Outcome: Cardiac Death or Myocardial Infarction (MI)
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 1.8 | 1.4

22. Secondary Outcome: Cardiac Death or Myocardial Infarction (MI)
Description: as for outcome 20
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 2.5 | 2.0

23. Secondary Outcome: All Death or Myocardial Infarction (MI)
Description: as for outcome 8
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 1.4 | 0.8

24. Secondary Outcome: All Death or Myocardial Infarction (MI)
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 2.0 | 1.7

25. Secondary Outcome: All Death or Myocardial Infarction (MI)
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 735
percentage of participants | 3.0 | 2.4

26. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: Target lesion revascularization is any ischemia-driven repeat percutaneous intervention to improve blood flow of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion.
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 0.8 | 0.1

27. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: TLR is any ischemia-driven repeat percutaneous intervention to improve blood flow of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 1.1 | 0.5

28. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 27
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 1.9 | 1.9

29. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: Target vessel revascularization is any ischemia-driven repeat percutaneous intervention to improve blood flow, or bypass surgery of not previously existing lesions with diameter stenosis ≥50% by quantitative coronary angiography in the target vessel, including the target lesion.
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 0.8 | 0.1

30. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: TVR is any ischemia-driven repeat percutaneous intervention to improve blood flow, or bypass surgery of not previously existing lesions with diameter stenosis ≥50% by quantitative coronary angiography in the target vessel, including the target lesion.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 1.2 | 0.7

31. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 30
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 2.9 | 2.7

32. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition
Description: DEFINITE ST: acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE ST: unexplained death within 30 days or target-vessel infarction without angiographic information ARC ST is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute ST: 0-24 hours after stent implantation; Subacute ST: >24 hours to 30 days post; late ST: >30 days to 1 year post; Very late ST: >1 year post; NOTE: Acute/subacute can be replaced by early ST (0-30 days).
Time Frame: 24 hours
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 762 | 768
percentage of participants | 0.1 | 0.1

33. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 32
Time Frame: >24 hr-30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 762 | 766
percentage of participants | 0.3 | 0.0

34. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 32
Time Frame: >30 days-1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 760 | 764
percentage of participants | 0.0 | 0.3

35. Secondary Outcome: Composite of All Death, All Myocardial Infarction (MI), All Target Vessel Revascularization (TVR)
Description: See above for definitions of MI and TVR
Time Frame: 30 days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 766
percentage of participants | 1.6 | 0.9

36. Secondary Outcome: Composite of All Death, All Myocardial Infarction (MI), All Target Vessel Revascularization (TVR)
Description: See above for definitions of MI and TVR.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 759 | 765
percentage of participants | 2.4 | 2.4

37. Secondary Outcome: Composite of All Death, All Myocardial Infarction (MI), All Target Vessel Revascularization (TVR)
Description: See above for definitions of MI and TVR.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 732 | 745
percentage of participants | 4.9 | 5.0

38. Secondary Outcome: Clinical Procedural Success
Description: Defined as mean lesion diameter stenosis <30% with visually assessed TIMI 3 flow and without the occurrence of in-hospital myocardial infarction (MI), target vessel revascularization (TVR), or cardiac death
Time Frame: In hospital
Population: Analysis was intention to treat (all patients in study).
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 761 | 767
percentage of participants | 98.2 | 98.3

39. Secondary Outcome: Acute Technical Success
Description: Defined as successful delivery and deployment of the study stent to the target vessel, without balloon rupture or stent embolization; expressed per stent
Time Frame: Acute-At time of index procedure
Population: Analysis was intention to treat (all patients in the study).
Measure: Number; unit: percentage of stents
Units Other Than Participants: Stents
Arm/Group | PROMUS | PROMUS Element
Number analyzed (Participants) | 762 | 768
Number analyzed (Stents) | 894 | 887
percentage of stents | 98.8 | 99.4

ADVERSE EVENTS:
Time Frame: Site reported other adverse events were collected through 365 days.
Arm/Group | PROMUS | PROMUS Element
Serious Adverse Events (participants affected / at risk) | 237/762 | 238/768
Other Adverse Events (participants affected / at risk) | 190/762 | 197/768
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS (N=762) | PROMUS Element (N=768)
Angina pectoris (Cardiac disorders) | 35 (39) | 44 (48)
Angina unstable (Cardiac disorders) | 9 (9) | 15 (17)
Coronary artery dissection (Cardiac disorders) | 14 (15) | 8 (8)
Coronary artery disease (Cardiac disorders) | 4 (5) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 4 (5)
Myocardial ischemia (Cardiac disorders) | 3 (3) | 5 (5)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (5)
Bradycardia (Cardiac disorders) | 4 (4) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery thrombosis (Cardiac disorders) | 3 (3) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 5 (6) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 4 (5) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy acute (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradychardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 32 (37) | 26 (28)
Chest pain (General disorders) | 8 (8) | 7 (7)
Catheter site haematoma (General disorders) | 1 (1) | 2 (2)
Adverse drug reaction (General disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Ulcer (Cardiac disorders) | 1 (1) | 0 (0)
Intermittant claudication (Vascular disorders) | 1 (1) | 4 (4)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 2 (4)
Femoral arterial stenosis (Vascular disorders) | 3 (3) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Aortic aneurysm (Vascular disorders) | 1 (1) | 3 (3)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Catheter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (2) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstruction airways disease (Infections and infestations) | 1 (1) | 0 (0)
Pneomonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperventillation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 4 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Inguinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (General disorders) | 1 (1) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 7 (7)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Acute leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pseudarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 3 (5)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 2 (2)
Presyncope (Nervous system disorders) | 2 (3) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (4) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 4 (5)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 2 (2) | 3 (3)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS (N=762) | PROMUS Element (N=768)
Angina pectoris (Cardiac disorders) | 79 (86) | 65 (73)
Myocardial infarction (Cardiac disorders) | 28 (28) | 41 (41)
Adverse drug reaction (General disorders) | 28 (28) | 40 (44)
Catheter site haematoma (General disorders) | 41 (41) | 41 (42)
Non-cardiac chest pain (General disorders) | 53 (59) | 49 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to Sponsor for review at least 45 days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.